CLINICAL TRIAL: NCT06955221
Title: Effect of US-guided Alcohol Sclerotherapy for Endometriomas on Pelvic Pain and Quality of Life
Brief Title: Effect of Alcohol Sclerotherapy on Pelvic Pain and Quality of Life in Women With Ovarian Endometriosis
Acronym: ESCOMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, Amparo Garcia-Tejedor, Clinical Professor, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR 070/25
Record Dates: First submitted 2025-04-08; First posted 2025-05-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Endometrioma; Ultrasound Therapy; Complications; Quality of Life; Pelvic Pain
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided aspiration and alcohol sclerotherapy (Experimental): US-guided alcohol sclerotherapy of endometriomas with absolute etanol during 15 minutes, followed by a posterior wash.
  Interventions: Procedure: Ultrasound-guided aspiration and alcohol sclerotherapy
- Control group (No Intervention): Expectant management with standard pain management if required

INTERVENTIONS:
Procedure: Ultrasound-guided aspiration and alcohol sclerotherapy — Ultrasound-guided puncture and alcohol sclerotherapy
  Arms: Ultrasound-guided aspiration and alcohol sclerotherapy

SUMMARY:
The goal of this clinical trial is to evaluate whether ultrasound-guided alcohol sclerotherapy can improve pelvic pain and quality of life in women aged 18 to 45 diagnosed with ovarian endometriomas, compared to expectant management.

The main questions it aims to answer are:

1. - Does sclerotherapy significantly reduce pelvic pain compared to expectant management?
2. - Does sclerotherapy improve quality of life as measured by the EHP-5 score?

Researchers will compare the sclerotherapy group to the expectant management group to determine whether the intervention leads to greater improvement in pain and quality of life.

Participants will:

* Be randomly assigned to one of two groups: (1) Sclerotherapy group: undergo ultrasound-guided puncture and alcohol sclerotherapy; (2) Control group: expectant management
* Complete quality of life and pain assessments at baseline and after 6 months
* Provide blood and urine samples for biomarker analysis (e.g., cortisol, IL-6, hsCRP, catecholamines)
* Undergo ovarian reserve assessments (AMH, antral follicle count)
* Be followed for adverse events, recurrence, fertility outcomes, and treatment-related costs

The study will follow an intention-to-treat and per-protocol analysis approach.

DETAILED DESCRIPTION:
Endometriosis is a chronic gynecological disease that affects women of reproductive age, characterized by the abnormal growth of endometrial tissue outside the uterine cavity.

It affects 5-10% of women of reproductive age (Becker et al., 2022) and is associated with infertility in 40% of cases (Coccia et al., 2008). Among its clinical forms, ovarian endometrioma is the most frequent, appearing in 15-45% of patients with endometriosis (Cranney et al., 2017). In addition to its impact on fertility, the main clinical manifestation of endometriosis is pain. Chronic pelvic pain caused by endometriosis can be disabling and even lead to work absenteeism, with a significant impact on the quality of life of affected patients, who often experience delayed diagnosis, making its management even more difficult and requiring a multidisciplinary approach (Horne & Missmer, 2022).

Currently, there is still no consensus on what should be the first-line treatment for ovarian endometrioma (Gordts & Campo, 2019). However, cystectomy reduces ovarian reserve due to the removal of healthy ovarian tissue adjacent to the cyst wall-something that further worsens the reproductive prognosis in patients whose fertility is already diminished due to endometriosis per se (Alborzi et al., 2021; Martinez-Garcia et al., 2021). Moreover, despite surgical removal of the endometrioma, the recurrence rate is high, ranging from 15-30% (Jee, 2022).

In recent years, there has been a shift toward more conservative treatments for the management of endometrioma, such as expectant management or aspiration and sclerosis (Garcia-Tejedor et al., 2020). Various authors have shown that ultrasound-guided aspiration and alcohol sclerosis may be a promising option, as concluded in the meta-analysis by Cohen et al., which found that recurrence rates were similar to those of laparoscopic management of ovarian endometrioma, but with fewer complications. Results in assisted reproductive technology are also better compared to surgical treatment in symptomatic women, particularly in those with low ovarian reserve (Zhang et al., 2022). Furthermore, other comparative studies between surgery and aspiration-sclerosis have shown that, although recurrence rates are similar, pregnancy rates are higher in patients treated with sclerosis, with the same complication rate and significantly lower costs (Garcia-Tejedor et al., 2020; Zhang et al., 2022).

Currently, the first-line treatment in patients diagnosed with endometriosis is hormonal therapy through the use of hormonal contraceptives. However, its efficacy in managing endometrioma is lower, and therefore, there is no consensus on its indication for this specific form of endometriosis (Cranney et al., 2017). In patients with a desire for pregnancy, alternative approaches are sought that do not interfere with fertility. At present, this often involves proceeding with in vitro fertilization without treating the endometrioma first, followed by surgery if needed (Miquel et al., 2020).

In addition to reproductive outcomes in patients affected by endometriosis, symptomatology and its consequent impact on quality of life have become highly relevant factors in treatment selection. Accordingly, specific pain scales and quality-of-life questionnaires have been developed to assess the impact on women affected by this condition. One such tool is the Endometriosis Health Profile scale, available in two versions (EHP-30 and EHP-5), designed by Dr. Stephen Kennedy and his team at the University of Oxford. It is a validated scale for assessing quality of life in patients with endometriosis and has been translated into nearly all languages (Jones et al., 2023; Bourdel et al., 2019).

The main objective of this project is to conduct a comparative analysis of patients diagnosed with ovarian endometrioma who undergo alcohol aspiration and sclerosis versus patients managed expectantly.

The outcomes to be evaluated include impact on quality of life, clinical improvement, pregnancy rate, and the need for subsequent surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age ≥18 and ≤45 years
* Ultrasound suspicion of unilocular endometrioma or with a thin septum less than 3 mm
* Size between 30-100 mm, persistent for at least 3-6 months since diagnosis
* Ca125 marker <300 UI/mL and HE4 < 70 pM
* Signed informed consent

Exclusion Criteria:

* Age <18 or >45 years
* History of ovarian or uterine cancer
* Endometrioma size <30 mm or >100 mm
* Indication for surgical treatment of the endometrioma due to suspected severe extra-ovarian endometriosis or any other cause
* Ultrasound suspicion of dermoid cysts, anechoic cysts, or cysts with high risk of malignancy
* Ca125 >300 UI/mL
* HE4 >70 pM
* Pregnant women
* Patients who do not wish to participate in the study or who are mentally incapacitated

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life of patients with endometrioma | Baseline and at 6 months
  Endometriosis Health Profile-5 (EHP-5), the minimum and maximum values (1-5), higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Pelvic pain | Baseline and at 6 months
  Visual Analog Score for pain (dysmenorrhea), the minimum and maximum values (0-10), higher scores mean a worse outcome.
Fertility preservation | Baseline and at 6 months
  Blood test: Antimullerian Hormone
Antral follicle | Baseline and at 6 months
  Antral follicle count by US
Pregnacy | through study completion, an average of 2 year
  Number of spontaneous pregnancies or pregnancies achieved through assisted reproductive techniques

CONTACTS AND LOCATIONS:
Overall Officials: Amparo Garcia-Tejedor, MDPhD, Principal Investigator — Hospital Universitari de Bellvitge; Rodrigo Javier Guevara-Peralta, Principal Investigator — Hospital Universitari de Bellvitge
Locations (26):
- Spain (26):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Consorci Sanitari de l'Anoia, Igualada, Barcelona
  - Consorci Sanitari Integral, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Consorci Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Parc Sanitari Sant Joan de Deu, Sant Boi de Llobregat, Barcelona
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital de Viladecans, Viladecans, Barcelona
  - Hospital Universitario Doctor José Molina Orosa, Arrecife, Canary Islands
  - Hospital Universitario San Pedro, Logroño, La Rioja
  - Hospital General Universitario Los Arcos del Mar Menor, San Javier, Murcia
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Joan XXIII, Tarragona
  - Hospital Recoletas Salud Campo Grande, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario de Álava - Txagorritxu, Vitoria-Gasteiz, Álava

IPD SHARING:
Plan to Share IPD: No